CLINICAL TRIAL: NCT04816175
Title: Intensive Therapy for Children With Microcephaly, Hyperkinetic Movements, or Global Developmental Delay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: American Academy of Cerebral Palsy and Developmental Medicine (Other)
Responsible Party: Principal Investigator, Stephanie DeLuca, Principal Investigator, Virginia Polytechnic Institute and State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #18-490
Record Dates: First submitted 2021-01-22; First posted 2021-03-25 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Microcephaly; Hyperkinesis With Developmental Delay; Global Developmental Delay
Keywords: Global Developmental Delay; Hyperkinesis; Microcephaly; Neurorehabilitation; Intensive Interventions
MeSH Terms: conditions — Microcephaly; Learning Disabilities; Hyperkinesis

STUDY DESIGN:
Intervention Model Description: As an early phase study, all enrolled children will receive the intervention.
Masking Description: Because all children will receive the intervention all parties involved will be aware that the participant has received the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Intervention (Experimental): All children will receive 3-5 weeks of intensive neuromotor Acquire therapy, an operant conditioning, play based therapy that maximizes therapeutic movements, attention, and engagement.
  Interventions: Behavioral: Acquire Therapy

INTERVENTIONS:
Behavioral: Acquire Therapy — This intervention is an operant conditioning based neurorehabilitation protocol for the promotion of psychomotor function

SUMMARY:
This trial will consist of a clinical series of up to 50 children with Global Developmental Delay and concomitant microcephaly or hyperkinetic movements. All children will be assessed for psychomotor function using standardized assessments, goal specific assessments, with the potential addition of neuroimaging assessment, prior to and after receiving an intensive burst of neuromotor therapy. The interventional effects will be explored by comparing the pre and post interventional assessments and neuroimaging.

DETAILED DESCRIPTION:
Up to 50 children between the ages of 6 months and 15 years will be recruited to participate in a burst of intensive neuromotor intervention in the form of Acquire therapy, delivered by the treatment team at Virginia Tech's Neuromotor Research Clinic. All children will have a diagnosis of Global Developmental Delay, with concomitant microcephaly or hyperkinetic movements. The children will be assessed for psychomotor function prior to and after the treatment intervention, using a series of standardized and goal specific assessments, with the possibility of additional neuroimaging assessments when possible. Acquire therapy is an intensive intervention in that it is delivered with high intensity, wherein goal directed behaviors are promoted at high levels of repetition and delivered at a high dose (4-6 hours a day) in an intensive burst of 3-4 weeks of 5 day a week treatment. Acquire therapy is an operant conditioning based intervention delivered in a cycle of refinement, reinforcement and repetition. It is play-based with activities selected to drive behavior toward goals that are specific to each child and selected based on each child's interests and needs. As such a specific protocol cannot be outlined. However, all goal directed activities are designed to promote awareness of and engagement with others and the environment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Global Developmental Delay with Microcephaly or hyperkinetic movements.

Exclusion Criteria:

* Medical Instability
* Under 6 months of age over 15 years of age

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline on Motor Function Assessment | 5-12 weeks
  A validated motor function assessment tool the CanChild Gross Motor Function Measure -88 will be used to measure change on motor function. The child can score between 0 and 264 points. The higher the child's score the more tasks they were able to attempt and/or complete.

SECONDARY OUTCOMES:
Change from baseline on measure of EEG coherence in alpha band | 5-12 weeks
  EEG data will be analyzed for changes in coherence in alpha band. Pre and post coherence in alpha band will be probed for changes by electrode pair.
Change from baseline on measure of EEG coherence in theta band. | 5-12 weeks
  EEG data will be analyzed for changes in coherence in theta band. Pre and post coherence in theta band will be probed for changes by electrode pair.
Change from baseline on measure of EEG coherence in beta band. | 5-12 weeks
  EEG data will be analyzed for changes in coherence in beta band. Pre and post coherence in beta band will be probed for changes by electrode pair.
Change from baseline on measure of EEG coherence in delta band. | 5-12 weeks
  EEG data will be analyzed for changes in coherence in delta band. Pre and post coherence in delta band will be probed for changes by electrode pair.
Change from baseline on EEG power in alpha band. | 5-12 weeks
  EEG data will be analyzed for changes in power in alpha band. Pre and post power will be compared for alpha band.
Change from baseline on EEG power in beta band. | 5-12 weeks
  EEG data will be analyzed for changes in power in beta bands. Pre and post power will be compared for beta band.
Change from baseline on EEG power in theta band. | 5-12 weeks
  EEG data will be analyzed for changes in power in theta band. Pre and post power will be compared for theta band.
Change from baseline on EEG power in delta bands. | 5-12 weeks
  EEG data will be analyzed for changes in power in delta bands. Pre and post power will be compared for delta band.
Change from baseline on Disability Assessment | 5-12 weeks
  Using the Pediatric evaluation of disability inventory with scores ranging from 0-100 with higher scored indicating greater functionality.
Change from baseline on fMRI measures of connectivity | 5-12 weeks
  fMRI data will be probed for change from baseline on measures of connectivity.
Change from baseline on fMRI regional activation patterns. | 5-12 weeks
  fMRI data will be probed for change from baseline on measures of regional activation.
Change from baseline on Motor Assessment | 5-12 weeks
  Using the Peabody Developmental Motor Scales, the Peabody consists of 6 subtests, that are each completed according to the child's age as a starting point. If a child were to complete all 6 subtests, and were to start at the earliest age block for all subtests the child would complete 255 items, with scores ranging from 0-510, the higher the score the more tasks the child was able to complete.
Change from baseline on goal specific assessment | 5-12 weeks
  Using a goal specific assessment form developed in the neuromotor research clinic children will be assessed for changes on child specific goals using a metric goal attainment assessment method (See Mann, J 2020 Dev Neurorehab). The child will be measured on their percent change on child-specific goals, with ranges from 0 percent change to infinity percent change. The higher the percent change the more the child changed on that particular goal.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie C DeLuca, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Fralin Biomedical Research Institute at Virginia Tech, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeLuca SC, Wallace DA, Trucks MR, Mukherjee K. A clinical series using intensive neurorehabilitation to promote functional motor and cognitive skills in three girls with CASK mutation. BMC Res Notes. 2017 Dec 19;10(1):743. doi: 10.1186/s13104-017-3065-z. PMID 29258560
- [Background] Mann J, Wallace DA, DeLuca S. Case study on the use of intensive pediatric neurorehabilitation in the treatment of kernicterus. J Clin Mov Disord. 2020 Feb 3;7:1. doi: 10.1186/s40734-020-0084-z. eCollection 2020. PMID 32042435
- [Background] Ramey SL, DeLuca S, Stevenson RD, Case-Smith J, Darragh A, Conaway M. Children with Hemiparesis Arm and Movement Project (CHAMP): protocol for a multisite comparative efficacy trial of paediatric constraint-induced movement therapy (CIMT) testing effects of dosage and type of constraint for children with hemiparetic cerebral palsy. BMJ Open. 2019 Jan 15;9(1):e023285. doi: 10.1136/bmjopen-2018-023285. PMID 30782701